CLINICAL TRIAL: NCT00803283
Title: A Randomized, Open-Labeled, Multi-Center Study to Investigate the Safety and Efficacy of OROS Hydromorphone HCl Comparing With Morphine SR in Cancer Pain Patients
Brief Title: A Study to Compare Safety and Efficacy of Osmotic Release Oral Syytem (OROS) Hydromorphone Hydrochloride (HCl) With Morphine Sustain Release (SR) in Participants With Cancer Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015328; 42801PAI3008
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Cancer Pain
Keywords: Pain; Hydromorphone hydrochloride OROS; Morphine
MeSH Terms: conditions — Cancer Pain; Pain

ARMS (2):
- Hydromprphone Hydrochloride (HCl) OROS (Experimental): Participants will receive hydromorphone HCl OROS 8 milligram (mg) every 24 hours, for 3 to 14 days of titration phase. Hydromorphone HCl OROS will be continued as per Investigator's discretion for next 14 days of maintenance phase.
  Interventions: Drug: Hydromprphone Hydrochloride (HCl) OROS
- Morphine Sustain Release (SR) (Active Comparator): Participants will receive morphine SR 8 mg every 24 hours, for 3 to14 days of titration phase. Morphine SR will be continued as per Investigator's discretion for next 14 days of maintenance phase.
  Interventions: Drug: Morphine Sustain Release (SR)

INTERVENTIONS:
Drug: Hydromprphone Hydrochloride (HCl) OROS — Participants will receive hydromorphone HCl OROS 8 milligram (mg) every 24 hours, for 3 to 14 days of titration phase. Hydromorphone HCl OROS will be continued as per Investigator's discretion for next 14 days of maintenance phase.
  Arms: Hydromprphone Hydrochloride (HCl) OROS
Drug: Morphine Sustain Release (SR) — Participants will receive morphine SR 8 mg every24 hours, for 3 to14 days of titration phase. Morphine SR will be continued as per Investigator's discretion for next 14 days of maintenance phase.
  Arms: Morphine Sustain Release (SR)

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Osmotic Release Oral System (OROS) hydromorohone Hydrochloride (HCl) compared with morphine sustain release (SR) in participants with chronic (lasting a long time) malignant (cancerous) cancer pain.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (when more than 1 hospital or medical school team work on a medical research study), active-controlled, randomized (the study drug is assigned by chance) study to evaluate safety and efficacy of OROS extended-release (ER) hydromorhone HCl compared to twice daily morphine SR, in Taiwan participants with cancer pain. The study consists of 3 phases: Screening phase (14 days before administration of study drug), Dose titration phase (3 to 14 days) and Dose maintenance phase (14 days). This study will include 8 visits (Visit 1 [Day 1], Visit 2 [Day 1-13 telephonic], Visit 3 [Day 14], Visit 4 [Day 15 to Day 21 telephonic], Visit 5 [Day 22], Visit 6 [Day 23 to 27 telephonic] and Visit 7 [Day 28]). In dose titration phase, participants will be randomly assigned to 1 of the 2 treatments, OROS hydromorphone or morphine SR and dose of study medication will be adjusted every 48 hours at Investigator's discretion according to participant's analgesic (drug used to control pain) requirements. Morphine HCl will be used as rescue medication (maintained at 3 doses per day or less) for breakthrough pain. Participants primarily will be evaluated for equivalence of efficacy using the "worst pain" item of the brief pain inventory (BPI). Participants' safety will be monitored throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cancer pain and experiencing inadequate pain control on or approaching Step 2 of the World Health Organisation (WHO) analgesic ladder
* Participants with pain scores greater than and equal to 4 on the average in the last 24 hours
* Participants requiring or are expected to require not more than 540 milligram of oral morphine or morphine equivalent every 24 hours for the management of chronic cancer pain
* Participants who can reasonably be expected to achieve stable dose of opioid study medication for the duration of the trial
* Participants who can reasonably be expected to achieve stable dose of opioid study medication for the duration of the trial

Exclusion Criteria:

* Participants with pure or predominantly neuropathic pain or pain of unknown origin (where a mechanism or physical cause cannot be identified)
* Participants with acute pain or who have pain on movement
* Participants who have received a fentanyl patch within the last 5 days
* Participants intolerant or hypersensitive to hydromorphone or other opioids agonists (chemical substance capable of activating a receptor to induce a full or partial response)
* Participants with recent past history (within the previous 5 years) or current history of drug abuse or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS): Participants received hydromorphone HCl OROS 8 milligram (mg) every 24 hours, for 3 to 14 days of titration phase. Hydromorphone HCl OROS was continued as per Investigator's discretion for next 14 days of maintenance phase.
- Morphine Sustain Release (SR): Participants received morphine SR 8 mg every 24 hours, for Day 3 to14 of titration phase. Morphine SR was continued as per Investigator's discretion for next 14 days of maintenance phase.
Period: Overall Study
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Number; unit: Participants]
  >=18 to <=40 years | 0 | 1 | 1
  >=41 to <=60 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) Questionnaire Item 3 "Worst Pain" Score at Day 14
Description: The BPI is a questionnaire designed to assess the severity and impact of pain on quality of life. Total score ranges from 0=no pain to 10=extreme pain. BPI Questionnaire Item 3 "Worst Pain" will be assessed using the BPI questionnaire, score ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Day 14
Population: Study was terminated due to poor enrollment and no efficacy data were summarized due to very low sample size. Only safety data were summarized.
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: BPI Questionnaire Item 3 "Worst Pain" Score at Day 28
Description: as for outcome 1
Time Frame: Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: BPI Questionnaire Item 6 "How Much Pain You Have Right Now" Score
Description: The BPI is a questionnaire designed to assess the severity and impact of pain on quality of life. Total score ranges from 0=no pain to 10=extreme pain. BPI questionnaire Item 6 "how much pain you have right now" will be assessed using the BPI questionnaire, score ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, Day 14, Day 22 and Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: BPI Questionnaire Item "Pain Intensity" Score
Description: The BPI is a questionnaire designed to assess the severity and impact of pain on quality of life. Total score ranges from 0=no pain to 10=extreme pain. BPI questionnaire Item "Pain Intensity" will be assessed using the BPI questionnaire, score ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, Day 14, Day 22 and Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: BPI Questionnaire Item "Pain Relief" Score
Description: The BPI is a questionnaire designed to assess the severity and impact of pain on quality of life. Total score ranges from 0=no pain to 10=extreme pain. BPI questionnaire Item "Pain Relief" will be assessed using the BPI questionnaire. Pain relief was rated on a scale ranging from 0% (no relief) to 100% (complete relief).
Time Frame: Baseline, Day 14, Day 22 and Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: BPI Questionnaire Item "Pain Interference" Score
Description: The BPI is a questionnaire designed to assess the severity and impact of pain on quality of life. Total score ranges from 0=no pain to 10=extreme pain. BPI questionnaire Item "Pain Interference" will be assessed using the BPI questionnaire. Pain interference of general activity, mood, walking ability, normal work, relationships with others, sleep, and enjoyment of life will be rated on a scale ranging from 0 (no interference) to 10 (complete interference).
Time Frame: Baseline, Day 14, Day 22 and Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Patient's Global Assessment on Effectiveness
Description: Participants will evaluate effectiveness by providing rating on the question "'what is your rating of the overall effectiveness of the study medication during the titration or maintenance phase" using 5-point scale ranging from 1 to 5, where 1=poor,. 2=fair, 3=good, 4=very good and 5=excellent.
Time Frame: Day 14, Day 22 and Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Investigator's Global Assessment on Effectiveness
Description: Investigator will evaluate effectiveness by providing rating on the question "'what is your rating of the overall effectiveness of the study medication during the titration or maintenance phase" using 5-point scale ranging from 1 to 5, where 1=poor,. 2=fair, 3=good, 4=very good and 5=excellent.
Time Frame: Day 14, Day 22 and Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Times the Pain Medication Required for Breakthrough Pain
Description: The requirement of breakthrough pain medication will be recorded by participants. Morphine HCl, 10 mg, will be used as rescue medication for breakthrough pain.
Time Frame: Baseline up to Day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Mean Total Daily Dose (TDD) of Study Medication
Description: Mean total daily dose of study medication taken during study will be recorded by participants.
Time Frame: Baseline up to day 28
Population: as for outcome 1
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Arm/Group | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) | Morphine Sustain Release (SR)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone Hydrochloride (HCl) Oral Osmotic System (OROS) (N=1) | Morphine Sustain Release (SR) (N=1)
Oedema peripheral (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Chest discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study had inadequate number of participants. 'The study was terminated early and the data for efficacy assessments were missing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less